CLINICAL TRIAL: NCT02233530
Title: Identification and Intervention for Dementia in Elderly Africans (IDEA) Study: CST Trial
Brief Title: IDEA Study Cognitive Stimulation Therapy (CST) Trial in Nigeria
Acronym: IDEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Keith Gray (Other)
Collaborators: Grand Challenges Canada (Other); University of Ibadan (Other); Kilimanjaro Christian Medical Centre, Tanzania (Other); Newcastle University (Other); Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, William Keith Gray, Dr Willliam Gray, Northumbria Healthcare NHS Foundation Trust
Organization: Northumbria Healthcare NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IDEA_NIGERIA_CST1
Record Dates: First submitted 2014-08-30; First posted 2014-09-08 (Estimated); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-05

CONDITIONS: Dementia
Keywords: Dementia; Cognitive Stimulation Therapy; Quality of life; Cognitive impairment; Africa; Tanzania; Nigeria; Low- and Middle-income countries; Non-pharmacological intervention; Task-shifting; Cognitive screening
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CST intervention (Experimental): Outcomes at baseline will be compared with those immediately post intervention and at four weeks post-intervention.
  In accordance with the CST manual protocol, patients will be allocated to groups to ensure a spread of abilities and ensure inclusivity. No group contains only one individual of a particular religion or gender, such that they may feel left out. The investigators will allocate patients to groups to avoid excessive travel to the group meeting place, participants may be allocated to a group based on their geographical location. Individuals will be allocated to groups based on religion, gender and geographical location.
  Interventions: Behavioral: CST intervention

INTERVENTIONS:
Behavioral: CST intervention — The CST intervention comprises 14 sessions lasting 1-2 hours across 7 weeks. The CST manual has been adapted for use in this setting by members of our study team. Each session has a theme. Activities include tasks aimed at engaging participants in cognitive and physical tasks designed to improve quality of life. Sessions will be led and facilitated by a study nurse or occupational therapist. The sessions will be held at a local health centre of village hall.

SUMMARY:
This trials of cognitive stimulation therapy (CST) in Tanzania is part of the larger Identification and Intervention for Dementia in Elderly Africans (IDEA) study.

The overall aim of the IDEA study is to set up and evaluate sustainable programmes to facilitate diagnosis of, and therapy for, people with dementia led by local communities in sub-Saharan Africa. The investigators seek to improve quality of life for people with dementia and their caregivers.

Within this trial of CST, the investigators hypothesise that CST can significantly improve the quality of people with dementia and their carers living in Africa

DETAILED DESCRIPTION:
The project will address three specific challenges: 1) Integrate screening and core packages of services into routine primary health care. 2) Provide effective and affordable community-based care and rehabilitation. 3) Develop effective treatment for use by non-specialists, including lay healthcare workers with minimal training.

Dementia is under-diagnosed in sub-Saharan Africa (SSA) and treatment is rarely accessed or available. The burden of dementia on caregivers is high, with loss of income, and psychosocial stress common. However, large scale screening for dementia in such a setting is neither affordable nor sustainable. The purpose of this 3 year project is to provide a sustainable mechanism for diagnosis and therapeutic intervention for people with dementia. The investigators will use 2 complimentary, rural study sites, 1 in Nigeria, West Africa and 2 in Tanzania, East Africa. As a consequence our results should be generalizable to all SSA. Our approach is inexpensive and will have applicability to other low- and middle-income countries.

During Phase I the investigators will validate a screening tool, previously developed by members of our study team from data collected in Tanzania, and carry out a pilot study of the benefits of cognitive stimulation therapy (CST) when used in SSA for those already identified with dementia. During both of these activities the investigators will initiate training of local healthcare workers in diagnosis and management of people with dementia. In Phase II the investigators will engage with local communities to raise awareness of dementia. Building on previous work at both study sites, the investigators will initiate poster, newspaper and radio advertising and use mobile phone text messaging services (for relevant healthcare personnel) to increase awareness of the need to diagnose and intervene at an early stage. The investigators will empower local private pharmacies to help identify people with dementia, a relationship which will ultimately be mutually beneficial through the supply of medicines to treat risk factors for dementia, such as hypertension. The investigators will engage with local community leaders and government officials to assist us in this awareness raising, an approach that has proven successful in previous studies by our team in SSA. One of our study team (Dr Mushi (DM)) is a social scientist based in Tanzania and during Phase II the investigators will conduct qualitative research into attitudes and beliefs surrounding dementia and identify any barriers to diagnosis in both sites. The results of this research will be fed back to inform other phases of the study. Finally, in phase III the investigators will initiate a program of community based CST led by local occupational therapists (OTs) and nurse specialists. OTs and nurses will train caregivers in CST techniques and the investigators hope that the training will ultimately be led by caregivers allowing such therapy to become sustainable within communities in the longer term. The investigators will evaluate changes in cognition in people with dementia, and quality of life (QOL) in both people with dementia and their caregivers, post-intervention. The investigators will carry out a full economic evaluation of the effect of our program, to be led by a heath economist based at Newcastle University, United Kingdom.

This protocol cover the CST trial (Phase III of the study) in Nigeria

ELIGIBILITY:
Inclusion Criteria:

* Anyone with dementia living within the study site

Exclusion Criteria:

* The participant and the family should have consented to take part in the study.
* Unable to travel to the centre where the CST sessions will be held due to physical impairment (e.g. bedbound or immobile)
* After assessment by the study doctor, deemed unable to engage in CST sessions (e.g. follow instructions and participate in activities) due to severe physical or cognitive impairment.
* Profound deafness
* Total blindness
* Aphasia - they should be able to understand verbal communication and communicate verbally (mild impairments are acceptable).
* The participant should be able to sit in a group setting for 1 hour.
* There should not be agitation, depression or psychosis to an extent that the person would not be able to tolerate spending time with other people in a group setting

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adesola Ogunniyi, MD, Principal Investigator — University of Ibadan, Nigeria; Akin Adebiyi, Study Director — University of Ibadan
Locations (1):
- Lalupon, Lalupon, Oyo State, Nigeria

REFERENCES:
- [Background] Gray WK, Paddick SM, Kisoli A, Dotchin CL, Longdon AR, Chaote P, Samuel M, Jusabani AM, Walker RW. Development and Validation of the Identification and Intervention for Dementia in Elderly Africans (IDEA) Study Dementia Screening Instrument. J Geriatr Psychiatry Neurol. 2014 Jun;27(2):110-8. doi: 10.1177/0891988714522695. Epub 2014 Feb 26. PMID 24578459

RESULTS

PARTICIPANT FLOW:
Groups:
- CST Intervention: Outcomes at baseline will be compared with those immediately post intervention and at four weeks post-intervention.
  In accordance with the CST manual protocol, patients will be allocated to groups to ensure a spread of abilities and ensure inclusivity. No group contains only one individual of a particular religion or gender, such that they may feel left out. The investigators will allocate patients to groups to avoid excessive travel to the group meeting place, participants may be allocated to a group based on their geographical location. Individuals will be allocated to groups based on religion, gender and geographical location.
  CST intervention: The CST intervention comprises 14 sessions lasting 1-2 hours across 7 weeks. The CST manual has been adapted for use in this setting by members of our study team. Each session has a theme. Activities include tasks aimed at engaging participants in cognitive and physical tasks designed to improve quality of life. Sessions will be led and facilitated by a study nurse or occupational therapist. The sessions will be held at a local health centre of village hall.
Period: Overall Study
Arm/Group | CST Intervention
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Cognitive stimulation therapy participants. Participant received two sessions per week for seven weeks, with 14 sessions in total. Each session lasted between 45 and 60 minutes.
Arm/Group | Intervention
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants] — Age was recorded in years
  Participants
    <=18 years | 0
    Between 18 and 65 years | 0
    >=65 years | 9
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 81 [79 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Nigeria | 9

OUTCOME MEASURES:

1. Primary Outcome: World Health Organization Brief Quality of Life Measure (WHOQOL-Bref)
Description: Quality of life assessment in patients and carers. The minimum score is 4 and the maximum 20, with a higher score signifying better quality of life.
Time Frame: Baseline
Population: All baseline participants
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Intervention: Intervention group
Arm/Group | Intervention
Number analyzed (Participants) | 9
units on a scale | 10.3 [9.4 to 12.9]

2. Primary Outcome: World Health Organization Brief Quality of Life Measure (WHOQOL-Bref)
Description: as for outcome 1
Time Frame: An average of eight weeks from baseline
Population: All baseline participants
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 9
units on a scale | 14.9 [12.3 to 16.0]

3. Secondary Outcome: WHOQOL Bref
Description: as for outcome 1
Time Frame: An average of twelve weeks from baseline
Reporting Status: Not Posted

4. Secondary Outcome: IDEA Cognitive Screen
Description: Cognitive assessment in patients
Time Frame: Baseline
Reporting Status: Not Posted

5. Secondary Outcome: IDEA Cognitive Screen
Description: Cognitive assessment in patients
Time Frame: An average of eight weeks from baseline
Reporting Status: Not Posted

6. Secondary Outcome: IDEA Cognitive Screen
Description: Cognitive assessment in patients
Time Frame: An average of twelve weeks from baseline
Reporting Status: Not Posted

7. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: Anxiety and depression assessment in patients and carers. The minimum score is 0 and the maximum 42, with a higher score signifying greater depression.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 9
units on a scale | 21 [19 to 21.5]

8. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: as for outcome 7
Time Frame: An average of eight weeks from baseline
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 9
units on a scale | 20 [18.5 to 21]

9. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: Anxiety and depression assessment in patients and carers
Time Frame: An average of twelve weeks from baseline
Reporting Status: Not Posted

10. Secondary Outcome: Zarit Burden Interview (ZBI)
Description: Carer burden assessment. The minimum score is 0 and the maximum 48, with a higher score signifying greater carer burden.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 9
units on a scale | 18 [10 to 35.5]

11. Secondary Outcome: Zarit Burden Interview (ZBI)
Description: Carer burden assessment. The minimum score is 0 and the maximum 48, with a higher score signifying greater carer burden.
Time Frame: An average of eight weeks from baseline
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 9
units on a scale | 11 [7.5 to 18]

12. Secondary Outcome: Zarit Burden Interview (ZBI)
Description: Carer burden assessment
Time Frame: An average of twelve weeks from baseline
Reporting Status: Not Posted

13. Secondary Outcome: Adapted Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog)
Description: Cognitive assessment in patients. The minimum score is 0 and the maximum 70, with a lower score signifying better cognition.
Time Frame: Baseline
Measure: Least Squares Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 9
units on a scale | 12 [5.5 to 35.5]

14. Secondary Outcome: Adapted Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog)
Description: as for outcome 13
Time Frame: An average of eight weeks from baseline
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 9
units on a scale | 7 [3.5 to 10.5]

15. Secondary Outcome: Adapted Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog)
Description: Cognitive assessment in patients
Time Frame: An average of twelve weeks from baseline
Reporting Status: Not Posted

16. Secondary Outcome: Study Specific Economic Evaluation
Description: Assessment of health service utilisation and time and travel for patients and carers
Time Frame: Baseline
Reporting Status: Not Posted

17. Secondary Outcome: Study Specific Economic Evaluation
Description: Assessment of health service utilisation and time and travel for patients and carers
Time Frame: An average of twelve weeks from baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During the intervention
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No